CLINICAL TRIAL: NCT04995406
Title: Validating the Use of Blood Transcriptomic Signatures for the Diagnosis of Active Pulmonary Tuberculosis With the ISIT-TB Prototype in Adults Living in a High Burden Setting
Brief Title: Validating the Use of Blood Transcriptomic Signatures for the Diagnosis of Active Pulmonary Tuberculosis
Acronym: ISIT-TB
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: ISIT-TB 001
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: TUBERCULOSIS, PULMONARY
Keywords: Tuberculosis; Mycobacterium infections; Bacterial infections; Diagnosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Mycobacterium Infections; Bacterial Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Active TB ATB: Participants with active tuberculosis with diagnosis confirmed by GeneXpert and/or culture positivity
  Interventions: Diagnostic Test: ISIT-TB prototype
- Latent Tuberculosis Infections LTBI: Participants with presumed latent TB infection
  Interventions: Diagnostic Test: ISIT-TB prototype
- Healthy controls HC: Participants who do not have Active or Latent tuberculosis or other pathologies investigated in this study
  Interventions: Diagnostic Test: ISIT-TB prototype
- Non-tuberculous symptomatic participants: This cohort refers to participants who are known with chronic respiratory conditions and present with one or more signs and symptoms suggestive of TB, but in whom microbiological testing is negative.
  Interventions: Diagnostic Test: ISIT-TB prototype

INTERVENTIONS:
Diagnostic Test: ISIT-TB prototype — Diagnostic assay able to identify active tuberculosis using a patient blood sample processed on an automatized system within an hour

SUMMARY:
ISIT-TB Prototype is a diagnostic assay based on a transcriptional blood signature suggestive of the detection of Mycobacterium tuberculosis.

DETAILED DESCRIPTION:
This device will be investigated for use as a screening tool to facilitate diagnosis of ATB in conjunction with risk assessment, clinical context and diagnostic information. Whole blood samples will be collected in Tempus™ Blood RNA Tubes and processed on an automatized platform. The detection of a combination of under or over-expressed selected genes, constituting a transcriptional signature, will allow the characterization of ATB.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggestive of TB disease: cough for more than two weeks plus at least one of the following: fever, malaise, weight loss, night sweats, haemoptysis, chest pain or loss of appetite.
* Willingness to give consent to take part in the study.
* Aged >18 years old.
* Healthy control : no history of TB treatment, no respiratory symptoms, no evidence of active infectious disease, no history of close contacts of active pulmonary TB patients.

Exclusion Criteria:

* Pregnant woman
* A person who has received treatment for active TB or LTBI in the past 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active TB cases will be prospectively recruited from the primary care TB clinics and participating hospitals. Healthy adults will be recruited using the healthy participant database of the participating hospitals. For LTBI population, individuals presenting to primary care facilities for reasons other than suspected TB will be approached and invited to participate as possible LTBI should they be assessed as being at increased risk for TB infection as described in the inclusion/exclusion criteria. Non-infectious respiratory disease controls will be recruited from the participing hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of performance of the diagnostic tool | Time to bacteriological confirmation 60 days
  Determination of the specificity and sensitivity of the diagnostic assay ISIT-TB Prototype for TB in a population living in a high-burden country

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, Pr, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town Lung Institute, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No